CLINICAL TRIAL: NCT06593782
Title: A Multicenter, Randomized, Double-blind, Active-Controlled Dose-Finding Study of HSK21542 Injection for the Prevention of Chemotherapy-induced Nausea and Vomiting (CINV)
Brief Title: Evaluating the Efficacy and Safety of HSK21542 Injection in Chemotherapy-induced Nausea and Vomiting
Acronym: CINV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSK21542-501
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
MeSH Terms: conditions — Nausea; Vomiting | interventions — dolasetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK21542-A (Experimental)
  Interventions: Drug: HSK21542
- HSK21542-B (Experimental)
  Interventions: Drug: HSK21542
- Dolasetron (Active Comparator)
  Interventions: Drug: Dolasetron

INTERVENTIONS:
Drug: HSK21542 — 1. HSK21542 injection was administered day 1;
  2. Placebo to match Dorasetron was administered on day 1;
  3. Aprepitant injection was administered on day 1;
  4. Dexamethasone tablets was administered on day 1 to day 4;
  Arms: HSK21542-A
Drug: HSK21542 — 1. HSK21542 injection was administered day 1;
  2. Placebo to match Dorasetron was administered on day 1;
  3. Aprepitant injection was administered on day 1;
  4. Dexamethasone tablets was administered on day 1 to day 4;
  Arms: HSK21542-B
Drug: Dolasetron — 1. Placebo to match HSK21542 injection was administered day 1;
  2. Dorasetron injection was administered on day 1;
  3. Aprepitant injection was administered on day 1;
  4. Dexamethasone tablets was administered on day 1 to day 4;
  Arms: Dolasetron

SUMMARY:
This is a multicenter, randomized, double-blind, active-controlled dose-finding study. About 180 subjects who receive a high emetic chemotherapy are planned to be enrolled and randomized into three groups by a ratio of 1:1:1.

ELIGIBILITY:
Inclusion Criteria:

1.18 years of age or older, of either gender;

2. Has never been treated with chemotherapy regimen and plan to receive asingle day high emetic chemotherapy regimen by intravenous infusion，including but not limited to AC regimen, carboplatin AUC ≥ 4, Camustine&gt;250 mg/m2, cisplatin, and other treatment options;

3. Diagnosed with a malignant solid tumor by histology or cytology;

4. Has an ECOG Performance Status of 0 or 1;

5. Predicted life expectancy of ≥3 months;

6. Adequate bone marrow, kidney, and liver function:

1. Absolute neutrophil count ≥ 1.5 × 109/L, white blood cell count ≥ 3.0 × 109/L;
2. Platelet count ≥ 75 × 109/L;
3. Hemoglobin ≥ 70 g/L;
4. Aspartate transaminase (AST) ≤ 3 × ULN (≤ 5 × ULN in patients with hepatocellular carcinoma or liver metastasis);
5. Alanine transaminase (ALT) ≤ 3 × ULN (≤ 5 × ULN in patients with hepatocellular carcinoma or liver metastasis);
6. Serum total bilirubin ≤ 2 × ULN (≤ 3 × ULN for patients with hepatocellular carcinoma or liver metastasis);
7. Creatinine ≤ 2 × ULN;

   7. Subjects who agree to participate in the trial and voluntarily sign the Informed Consent Form (ICF);

Exclusion Criteria:

1. History or evidence of any of the following diseases prior to screening:

   1. Suffering from primary or metastatic malignant tumors of the central nervous system;
   2. Suffering from epilepsy, Parkinson&amp;amp;#39;s disease, or other central nervous system disorders that cause nausea and vomiting;
   3. Suffering from intestinal obstruction or other digestive system diseases that may cause nausea and vomiting as determined by researchers;
   4. Suffering from clearly diagnosed vestibular dysfunction other than motion sickness (including but not limited to peripheral vestibular syndrome, central vestibular syndrome, etc.);
   5. History of obvious and chronic dizziness;
   6. QT interval&amp;amp;gt;450 ms during screening or taking concomitant medications due to prolonged QT interval or has risk factors for QT interval prolongation or correspon;
2. Allergies or contraindications to the study drugs or other drugs specified in the protocol (including chemotherapy drugs, investigational drugs and mimetics, dorasetron, aripipitan, dexamethasone, etc.) ;
3. Subjects who have experienced nausea, retching, or vomiting before 24 hours of randomization;
4. Subjects who have received abdominal or pelvic radiation therapy within the first 7 days of randomization or plan to receive abdominal or pelvic radiation therapy during the study period;
5. Subjects with a history of drug abuse, drug addiction, or alcoholism within 3 months prior to screening, where alcoholism is defined as consuming >2 units of alcohol on average daily (1 unit = 360 mL of beer with 5% alcohol, 45 mL of liquor with 40% alcohol or 150 mL of wine);
6. Subjects who have participated in any investigational trial (defined as receiving investigational drug or placebo) within 1 month prior to screening;
7. Female subjects who are pregnant or breastfeeding; female or male subjects of child-bearing potential are unwilling to use contraception throughout the entire study period and for 3 months after the study completion;
8. Subjects judged by the investigator to be unsuitable for participating in this clinical trial for any other factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-16 (Estimated); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Acute Complete response | 0 to 24 hours
  Acute Complete response was defined as no vomiting/retching and no rescue therapy over the first 24 hours after the initiation of high emetic chemotherapy regimen

SECONDARY OUTCOMES:
Overall Complete response | 0 to 120 hours
  Overall Complete response was defined as no vomiting/retching and no rescue therapy over the first 120 hours after the initiation of high emetic chemotherapy regimen
Delayed Complete response | 24 to 120 hours
  Delayed Complete response was defined as no vomiting/retching and no rescue therapy over the 24 to 120 hours after the initiation of high emetic chemotherapy regimen